CLINICAL TRIAL: NCT05150821
Title: Impact of Covid-19 in the Emergency Department in a Tertiary Care Hospital, Nuremberg-Germany
Brief Title: Impact of Covid-19 in the Emergency Department
Status: Completed | Type: Observational
Sponsor: Dr. Panagiota Manava (Other)
Responsible Party: Sponsor-Investigator, Dr. Panagiota Manava, Dr. med. Panagiota Manava, MD, Principal Investigator, Paracelsus Medical University
Organization: Paracelsus Medical University (Other)
Other Study IDs: IC_2021_KNN
Record Dates: First submitted 2021-12-07; First posted 2021-12-09 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- experimental: patients during lockdown
- control group: patients before lockdown

SUMMARY:
To investigate the effects of lockdown in the Emergency Department in a tertiary health care hospital, Nuremberg, Germany.

DETAILED DESCRIPTION:
To investigate the effect of the first lockdown caused by the pandemic of Covid-19 in a tertiary health care hospital. Klinikum Nuremberg is one of the largest tertiary health care hospitals in Germany with two locations in Nuremberg. In the north department, around 150 outcome patients visit the Emergency Department every day.

During the pandemic in 2020 the capacities of the hospitals were saved for the patients with Covid-19. A decrease of patients presented in the ED was noticed. Controlling system and patient management provided the number of cases and correlated with the same period of time one year ago, before the pandemic.

For the classification of severity of diseases, different clinical diseases with severity scores were analyzed. Following diseases and scores were evaluated:

Pancreatitis -- > ranson score; ACS (acute coronary syndrome) --> Grace-Score; Pulmonary Embolism -- > sPESI (simplified Pulmonary Embolism Severity Index); Diverticulitis --> CDD (Classification of Diverticular Disease); Pneumonia -> crb65 (Confusion- Respiratory rate- Blood pressure- age ≥ 65 years);

ELIGIBILITY:
Inclusion Criteria:

Only patients who presented in the ED.

Exclusion Criteria:

none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: the study population will be patients of a teriary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 599 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
ranson score | through study completion, an average of 1 year
  clinical severity index of pancreatitis. Estimates mortality of patients with pancreatitis, based on initial and 48-hour lab values. Min. 0 - Max. 11 points.
Grace-Score | through study completion, an average of 1 year
  clinical severity index of ACS. Estimates admission untill 6 month mortality for patients with acute coronary syndrome. 108 points: low risk. Over 141-372 points: high risk.
sPESI | through study completion, an average of 1 year
  clinical severity index of pulmonary embolism. Predicts 30-day outcome of patients with pulmonary embolism. Min 0 points- max. 6 points
crb65 | through study completion, an average of 1 year
  The CRB-65-score is a clinical score that is used to estimate the severity of community-acquired pneumonias. The score corresponds to the statistical probability of patients dying because of pneumonia. Min 0 points - highest score 4 points.
CDD | through study completion, an average of 1 year
  clinical severity index of diverticulitis. Min 0 - max. 4

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Radiology and Nuclear Medicine, Nuremberg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hwee J, Chiew J, Sechachalam S. The Impact of Coronavirus Disease 2019 (COVID-19) on the Practice of Hand Surgery in Singapore. J Hand Surg Am. 2020 Jun;45(6):536-541. doi: 10.1016/j.jhsa.2020.04.023. Epub 2020 Apr 29. PMID 32387156
- [Background] Tam CF, Cheung KS, Lam S, Wong A, Yung A, Sze M, Fang J, Tse HF, Siu CW. Impact of coronavirus disease 2019 (COVID-19) outbreak on outcome of myocardial infarction in Hong Kong, China. Catheter Cardiovasc Interv. 2021 Feb 1;97(2):E194-E197. doi: 10.1002/ccd.28943. Epub 2020 May 5. PMID 32367683
- [Background] Wexner SD, Cortes-Guiral D, Gilshtein H, Kent I, Reymond MA. COVID-19: impact on colorectal surgery. Colorectal Dis. 2020 Jun;22(6):635-640. doi: 10.1111/codi.15112. Epub 2020 May 22. PMID 32359223
- [Background] Morgan C, Ahluwalia AK, Aframian A, Li L, Sun SNM. The impact of the novel coronavirus on trauma and orthopaedics in the UK. Br J Hosp Med (Lond). 2020 Apr 2;81(4):1-6. doi: 10.12968/hmed.2020.0137. Epub 2020 Apr 10. PMID 32343187
- [Background] Wang Y, Han W, Pan L, Wang C, Liu Y, Hu W, Zhou H, Zheng X. Impact of COVID-19 on blood centres in Zhejiang province China. Vox Sang. 2020 Aug;115(6):502-506. doi: 10.1111/vox.12931. Epub 2020 Apr 29. PMID 32347566